CLINICAL TRIAL: NCT01133548
Title: A Multiple Dose Pharmacokinetic and Comparative Bioavailability Study of Testosterone Absorption After Administration of 5 g Testosterone Gel 1.62% to the Upper Arms/Shoulders Using an Application Site Rotation or a Combination of Application Sites in Hypogonadal Males
Brief Title: Pharmacokinetic and Comparative Bioavailability Study of Testosterone Absorption After Administration of Testosterone Gel 1.62% to the Upper Arms/Shoulders Using an Application Site Rotation or a Combination of Application Sites in Hypogonadal Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S176.1.010
Record Dates: First submitted 2010-05-21; First posted 2010-05-31 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2011-06

CONDITIONS: Hypogonadism
Keywords: testosterone, hypogonadal, males
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Testosterone Gel 1.62%
  Interventions: Drug: Testosterone Gel 1.62%

INTERVENTIONS:
Drug: Testosterone Gel 1.62% — 5 grams administered using an application Site Rotation
Drug: Testosterone Gel 1.62% — 5 grams administered using an a combination of Application sites

SUMMARY:
To evaluate the pharmacokinetics and comparative bioavailability of Testosterone absorption in 36 Hypogonadal males after administration of 5 g Testosterone Gel 1.62% to the upper arms/shoulders using an application site rotation or a combination of application sites.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetics and comparative bioavailability of Testosterone absorption in 36 Hypogonadal males after administration of 5 g Testosterone Gel 1.62% to the upper arms/shoulders using an application site rotation or a combination of application sites.

ELIGIBILITY:
Inclusion Criteria

1. Hypogonadal males
2. Screening testosterone <300 ng/dL

Exclusion Criteria

1. Smokers
2. Previous history of or current or suspected prostate or breast cancer

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration observed (Cmax) | Up to 24 days
  Maximum plasma concentration observed (Cmax) of total testosterone, dihydrotestosterone, estradiol
Area Under the Plasma Concentration-time Curve (AUC) | Up to 24 days
  Area under the plasma concentration-time curve (AUC) of total testosterone, dihydrotestosterone, estradiol
Time of Cmax (Tmax) | Up to 24 days
  Time of Cmax (Tmax) of total testosterone, dihydrotestosterone, estradiol
Average Plasma Concentration observed (Cav) | Up to 24 days
  Average plasma concentration observed (Cav) of total testosterone, dihydrotestosterone, estradiol

SECONDARY OUTCOMES:
Application site evaluation based on the clinical evaluation of skin reactions grading scale | 24 days
Adverse events | 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael miller, PharmD, Study Director — Abbott

REFERENCES:
- [Result] Kaufman JM, Miller MG, Garwin JL, Fitzpatrick S, McWhirter C, Brennan JJ. Efficacy and safety study of 1.62% testosterone gel for the treatment of hypogonadal men. J Sex Med. 2011 Jul;8(7):2079-89. doi: 10.1111/j.1743-6109.2011.02265.x. Epub 2011 Apr 14. PMID 21492400